CLINICAL TRIAL: NCT01049555
Title: Contribution of Actigraphy and Recognition Video in Apathy Assessment of Alzheimer's Disease : Experimental Research
Acronym: 09-PP-06
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 09-PP-06
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Alzheimer's Disease
Keywords: alzheimer; apathy; actigraphy
MeSH Terms: conditions — Alzheimer Disease; Lethargy | interventions — Actigraphy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alzheimer and apathy (Other): Alzheimer's disease patients with apathy
  Interventions: Other: Actigraphy and video recording signal
- alzheimer without disease (Other): Alzheimer's disease patients without apathy
  Interventions: Other: Actigraphy and video recording signal
- Case control (Other): subject without apathy neither Alzheimer's disease
  Interventions: Other: Actigraphy and video recording signal

INTERVENTIONS:
Other: Actigraphy and video recording signal — Actigraphy and video recording signal during 1 hour

SUMMARY:
Neuropsychiatric symptoms form part of the clinical picture of Alzheimer's disease (AD) and other dementias. Irrespective of the severity of the disease, the most frequently encountered symptom is apathy. Apathy is increasingly diagnosed in patients with neurological and psychiatric conditions. Apathy is a disorder of motivation, defined as "the direction, intensity and persistence of goal-directed behaviour". Most of the current descriptions acknowledge this point and consider apathy in terms of a lack of goal-directed behaviour, cognition or emotion. The classical neuropsychiatric symptom assessments are subjective structured interview-based, using input from the caregiver and/or the patient. New technologies are likely to provide us with a more objective measure. An example is ambulatory actigraphy, consisting of a piezoelectric accelerometer designed to record arm movement in three dimensions.

The aim of the present study is to assess using actigraphy and video recording signal, AD patients with (n = 15) and without (n = 15) apathy and control subjects (n = 5) during an activity of daily living scenario .

ELIGIBILITY:
Inclusion Criteria:

* male or female, > 65 years ;
* Alzheimer's disease according to the NINCDS-ADRDA criteria (McKhann,Drachman et al. 1984) ;
* Mini Mental Test Examination (MMSE) > 20 ;
* no motor anomaly according to UPDRS III (tremblements, rigidité musculaire) ;
* no depression criteria according to DSM IV-R criteria ;
* patient with a cholinergic treatment at dose stable since 3 months ;
* patient with social insurance ;
* signature of informed consent.

Exclusion Criteria:

* neuropsychologics assessment impossible due to sensorial and disrupt ;
* prescription of psychotrop treatment (hypnotic, anxiolytic, antidepressant, antipsychotic) in the week previous actigraphy recording.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
assessment of motricity | one time point - at the only visit of protocol

SECONDARY OUTCOMES:
video recording | one time point - at the only visit of the protocol

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ROBERT, PU-PH, Principal Investigator — Nice University Hospital
Locations (1):
- Nice University Hospital, Nice, France